CLINICAL TRIAL: NCT05321069
Title: A Double Blind, Randomized, Placebo-controlled Trial Evaluating the Efficacy and Safety of BI 1015550 Over at Least 52 Weeks in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study to Find Out Whether BI 1015550 Improves Lung Function in People With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1305-0014; 2022-001091-34 (EudraCT Number)
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — BI 1015550

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nerandomilast 9 mg BID (Experimental): Participants received 9 mg film-coated nerandomilast tablets orally twice daily, with doses administered at least 12 hours apart, each taken with 250 mL of water.
  Interventions: Drug: BI 1015550
- Nerandomilast 18 mg BID (Experimental): Participants received 18 mg film-coated nerandomilast tablets orally twice daily, with doses administered at least 12 hours apart, each taken with 250 mL of water.
  Interventions: Drug: BI 1015550
- Placebo (Placebo Comparator): Participants received placebo matching 9 mg or 18 mg nerandomilast film-coated tablets orally twice daily, with doses given at least 12 hours apart and each taken with 250 mL of water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1015550 — Participants received film-coated nerandomilast tablets orally twice daily at doses of either 9 mg or 18 mg, with each dose administered at least 12 hours apart and taken with 250 mL of water.
  Other Names: Nerandomilast, JASCAYD®
  Arms: Nerandomilast 18 mg BID; Nerandomilast 9 mg BID
Drug: Placebo — Participants received placebo matching 9 mg or 18 mg nerandomilast film-coated tablets orally twice daily, with doses given at least 12 hours apart and each taken with 250 mL of water.
  Arms: Placebo

SUMMARY:
This study is open to adults with a lung disease called Idiopathic Pulmonary Fibrosis (IPF). People can join the study if they are 40 years or older. If they already take nintedanib or pirfenidone for their IPF, they can continue treatment throughout the study. The purpose of this study is to find out whether a medicine called BI 1015550 helps people with IPF.

Participants are put into 3 groups randomly, which means by chance. Participants in 2 groups take different doses of BI 1015550 as tablets twice a day. Participants in the placebo group take placebo tablets twice a day. Placebo tablets look like BI 1015550 tablets but do not contain any medicine.

Participants are in the study for up to two and a half years. During the first year, they visit the study site 10 times. Afterwards, they visit the study site every 3 months. The doctors regularly test participants' lung function. The results of the lung function tests are compared between the groups. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

1. Patients ≥40 years old at the time of signed informed consent.
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
3. Diagnosis of Idiopathic Pulmonary Fibrosis (IPF).
4. Patients may be either:

   * on a stable therapy* with nintedanib or pirfenidone for at least 12 weeks prior to Visit 1 and during screening and are planning to stay on this background treatment after randomization. Combination of nintedanib plus pirfenidone is not allowed. (*stable therapy is defined as the individually and general tolerated regimen of either nintedanib or pirfenidone (no dose changes) for at least 12 weeks).
   * not on a treatment with nintedanib or pirfenidone for at least 8 weeks prior to Visit 1 and during the screening period (e.g. either Antifibrotic (AF)-treatment naïve or previously discontinued) and do not plan to start or re-start antifibrotic treatment.
5. Forced Vital Capacity (FVC) ≥45% of predicted normal at Visit 1.
6. Diffusing Capacity (of Lung) for Carbon Monoxide (DLCO) ≥25% of predicted normal corrected for hemoglobin (Hb) at Visit 1.
7. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control. WOCBP taking oral contraceptives (OCs) also have to use one barrier method.

Exclusion criteria

1. Prebronchodilator Forced Expiratory Volume in 1 second (FEV1)/Forced vital capacity (FVC) <0.7 at Visit 1.
2. In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
3. Acute Idiopathic Pulmonary Fibrosis (IPF) exacerbation within 3 months prior to Visit 1 and/or during the screening period (investigator-determined).
4. Relevant chronic or acute infections including human immunodeficiency virus (HIV) and viral hepatitis.
5. Confirmed infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) not fully recovered according to investigator judgement within the 4 weeks prior to randomization (Visit 2).
6. Major surgery (major according to the investigator's assessment) performed within 6 weeks prior to Visit 2 or planned during the trial period, e.g. hip replacement. Registration on lung transplantation list would not be considered as planned major surgery.
7. Any documented active or suspected malignancy or history of malignancy within 5 years prior to Visit 1, except appropriately treated basal cell carcinoma of the skin, in situ squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
8. Aspartate aminotransferase (AST) or Alanine Aminotransferase (ALT) >2.5 x Upper limit of normal (ULN) or total Bilirubin >1.5 x ULN at Visit 1.

Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1177 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (334):
- United States (56):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Clinical Research Specialists LLC, Kissimmee, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Destin Pulmonary Critical Care, Santa Rosa Beach, Florida
  - Piedmont Healthcare-Atlanta-57055, Atlanta, Georgia
  - Evanston Hospital Pulmonary Clinic, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Louisville Pulmonary Care, Louisville, Kentucky
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Beaumont Health, Royal Oak, Michigan
  - Minnesota Lung Center and Sleep Institute, Edina, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Northern Westchester Hospital, Mount Kisco, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medicine-New York-59955, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Research Center-Winston-Salem-61365, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Health Honickman Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Clinical Trials Center of Middle Tennessee, LLC, Franklin, Tennessee
  - Vanderbilt University Medical Center - Vanderbilt Lung Institute at 100 Oaks, Nashville, Tennessee
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (7):
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Consultorios Médicos del Buen Ayre, Capital Federal
  - Instituto Ave Pulmo, Mar del Plata
  - INSARES, Mendoza
  - Centro Respiratorio de Quilmes, Quilmes
- Australia (12):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Lung Research Queensland, Chermside, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Lung Research Victoria, Footscray, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Trialswest, Spearwood, Western Australia
- Austria (7):
  - LKH Klagenfurt am Woerthersee, Klagenfurt
  - Krems University Hospital, Krems
  - Hospital Elisabethinen Linz, Linz
  - LKH Salzburg University Hospital, Salzburg
  - AKH - Medical University of Vienna, Vienna
  - Clinic Floridsdorf, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (7):
  - Ziekenhuis Netwerk Antwerpen (ZNA) - Campus Middelheim, Antwerp
  - ULB Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UNIV UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Brazil (8):
  - Serviços Medicos Respirar Sul Fluminense, Barra Mansa
  - Hospital das Clinicas da Universidade Federal de Minas Gerais (HCUFMG), Belo Horizonte,Minas Gerais
  - Edumed - Educacao e Saude SA, Curitiba
  - CLARE - Clinica de Pneumologia, Goiânia
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Instituto D´Or de Pesquisa e Ensino - Bahia, Salvador
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Hospital Alemao Oswaldo Cruz, São Paulo
- Canada (12):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Kelowna Respirology & Allergy Research, Kelowna, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital (Vancouver), Vancouver, British Columbia
  - Dr. Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Dr. Syed Anees Medicine Professional Corporation, Windsor, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - CIC Mauricie Inc., Trois-Rivières, Quebec
  - IUCPQ (Laval University), Québec
- Chile (2):
  - Instituto Nacional del Tórax, Providencia, Santiago de Chile
  - Centro de Investigación del Maule, Talca
- China (33):
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - NanFang Hosptial, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The First hospital of Jiaxing, Jiaxing
  - Jinhua Municipal Central Hospital, Jinhua
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Huadong Hospital affiliated to Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - China Shenyang Chest Hospital, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - People's Hospital of Sichuan Province, Sichuan
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital Affiliated Tongji Medical College Huazhong University of S & T, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Second Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
  - Yichang Central People's Hospital, Yichang
- University Hospital Dubrava, Zagreb, Croatia
- Denmark (3):
  - Aarhus University Hospital, Aarhus N
  - Herlev and Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense
- North Estonia Medical Centre Foundation, Tallinn, Tallinn, Estonia
- Finland (2):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - Oulun yliopistollinen keskussairaala, Oulu
- France (23):
  - HOP d'Angers, Angers
  - HOP Avicenne, Bobigny
  - HOP de la Cavale Blanche, Brest
  - HOP Louis Pradel, Bron
  - HOP CHU Caen, Caen
  - HOP François Mitterrand, Dijon
  - HOP Michallon, La Tronche
  - HOP Bicêtre, Le Kremlin-Bicêtre
  - INS Coeur Poumon, Lille
  - HOP Nord, Marseille
  - HOP Nord Laennec, Nantes
  - HOP Pasteur, Nice
  - HOP Paris Saint-Joseph, Paris
  - HOP Tenon, Paris
  - HOP Bichat, Paris
  - HOP Haut-Lévêque, Pessac
  - HOP Robert Debré, Reims
  - HOP Pontchaillou, Rennes
  - HOP Charles Nicolle, Rouen
  - HOP Civil, Strasbourg
  - HOP Foch, Suresnes
  - HOP Larrey, Toulouse
  - HOP Bretonneau, Tours
- Germany (21):
  - Velocity Clinical Research Germany GmbH, Ahrensburg, Ahrensburg
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Klinikum Region Hannover GmbH, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikum Konstanz, Konstanz
  - Klinikum der Universität München - Campus Großhadern, München
  - Klinikum Nürnberg, Nuremberg
  - Krankenhaus Bethanien gGmbH, Solingen
  - Helios Hanseklinikum Stralsund, Stralsund
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Petrus-Krankenhaus, Wuppertal
- Greece (3):
  - Hospital of Heraklion (PAGNI), Crete
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - Univ. Gen. Hosp. of Patras, Pátrai
- Hungary (2):
  - Koranyi National Institute For Pulmonolgy, Budapest
  - University of Debrecen Clinical Centre, Debrecen
- Connolly Hospital Blanchardstown, Dublin, Ireland
- Italy (11):
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - A. O. Universitaria Careggi, Florence
  - Ospedale Colonnello D Avanzo, Foggia
  - Ospedale G.B. Morgagni, Forlì
  - Ospedale Classificato San Giuseppe, Milan
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Pol. Universitario Tor Vergata, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - A.O.U. Senese, Siena
  - Ospedali Riuniti di Ancona, Torrette Di Ancona (Ancona)
- Japan (33):
  - Tosei General Hospital, Aichi, Seto
  - Fujita Health University Hospital, Aichi, Toyoake
  - Chiba University Hospital, Chiba, Chiba
  - IUHW Narita Hospital, Chiba, Narita
  - University of Fukui Hospital, Fukui, Yoshida-gun
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Fukuoka, Iizuka
  - Kurume University Hospital, Fukuoka, Kurume
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Tsuboi Hospital, Fukushima, Koriyama
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Kobe City Hospital Organization Kobe City Medical Center West Hospital, Hyogo, Kobe
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kindai University Hospital, Osaka, Osakasayama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Saitama Red Cross Hospital, Saitama, Saitama
  - Shimane University Hospital, Shimane, Izumo
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Tokushima University Hospital, Tokushima, Tokushima
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - Toranomon Hospital, Tokyo, Minato-ku
  - Kyorin University Hospital, Tokyo, Mitaka
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
  - National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Malaysia (4):
  - Hospital Sultan Idris Shah Serdang, Kajang
  - Institut Perubatan Respiratori, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Hospital Pulau Pinang-Pulau Pinang-21953, Pulau Pinang
- Mexico (5):
  - Centro de Investigacion Integral MEDIVEST S.C, Chihuahua City
  - Soltmed Smo, Mexico City
  - Centro Respiratorio de Mexico, Mexico City
  - Centro de Prevención y Rehabilitación de Enfermedades Pulmon, Monterrey
  - Oaxaca Site Management Organization, S.C., Oaxaca City
- Netherlands (3):
  - Zuyderland Medisch Centrum, Heerlen
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam
- New Zealand (4):
  - Waikato Hospital, Hamilton
  - Greenlane Clinical Centre, One Tree Hill, Auckland
  - Middlemore Clinical Trials, Papatoetoe
  - Tauranga Hospital, Tauranga South
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Akershus Universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Poland (3):
  - University Clinical Center, Gdansk, Gdansk
  - Alergopneuma Medical Center, Świdnik
  - Nat.Instit.of Tuberculosis&LungDiseases,Outpat.Clin,warszawa, Warsaw
- Portugal (2):
  - ULS de Coimbra, E.P.E., Coimbra
  - USLM, EPE - Hospital Pedro Hispano, Matosinhos Municipality
- Allianze Pulmonary Research LLC, Guaynabo, Puerto Rico
- Singapore (3):
  - National University Hospital-Singapore-42005, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Africa (3):
  - Busamed Paardevlei Private Hospital, Cape Town
  - Melomed Gatesville Hospital, Cape Town
  - KwaPhila Health Solutions, Durban
- South Korea (8):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (25):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital de Galdakao, Galdakao
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital General Universitario de Valencia, Valencia
- Sweden (3):
  - Universitetssjukhuset, Linköping, Linköping
  - Sahlgrenska Universitetsjukhuset, Stockholm
  - Akademiska sjukhuset, Uppsala
- Universitätsspital Basel, Basel, Switzerland
- Taiwan (6):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (6):
  - Siriraj Hospital, Bangkok Noi
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Khon Kaen
  - Central Chest Institute of Thailand, Muang
  - Maharat Nakhonchiangmai Hospital, Muang
  - Ramathibodi Hospital, Ratchatewi
- United Kingdom (9):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Southmead Hospital, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Royal Lancaster Infirmary, Lancaster
  - St James's University Hospital, Leeds
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Wuyts WA, Richeldi L, Assassi S, Azuma A, Cottin V, Hoffmann-Vold AM, Kreuter M, Oldham JM, Martinez FJ, Valenzuela C, Wijsenbeek MS, Kanakapura M, James A, Weimann G, Drzewuski C, Coeck C, Maher TM. Design of an open-label extension trial of nerandomilast (BI 1015550) in patients with idiopathic pulmonary fibrosis and progressive pulmonary fibrosis (FIBRONEER-ON). BMC Pulm Med. 2025 Dec 4;26(1):10. doi: 10.1186/s12890-025-03973-7. PMID 41345848
- [Derived] Richeldi L, Azuma A, Cottin V, Kreuter M, Maher TM, Martinez FJ, Oldham JM, Valenzuela C, Clerisme-Beaty E, Gordat M, Wachtlin D, Liu Y, Schlecker C, Stowasser S, Zoz DF, Wijsenbeek MS; FIBRONEER-IPF Trial Investigators. Nerandomilast in Patients with Idiopathic Pulmonary Fibrosis. N Engl J Med. 2025 Jun 12;392(22):2193-2202. doi: 10.1056/NEJMoa2414108. Epub 2025 May 18. PMID 40387033
- [Derived] Richeldi L, Azuma A, Cottin V, Kreuter M, Maher TM, Martinez FJ, Oldham JM, Valenzuela C, Gordat M, Liu Y, Stowasser S, Zoz DF, Wijsenbeek MS. Design of a phase III, double-blind, randomised, placebo-controlled trial of BI 1015550 in patients with idiopathic pulmonary fibrosis (FIBRONEER-IPF). BMJ Open Respir Res. 2023 Aug;10(1):e001563. doi: 10.1136/bmjresp-2022-001563. PMID 37597969
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled, multi-centre, Phase III trial evaluating the efficacy, safety, and tolerability of nerandomilast (BI 1015550) 9 mg and 18 mg bid versus placebo in patients with IPF. The trial included two parts: Treatment Period A lasted up to 52 weeks post-randomisation, followed by Treatment Period B with continued blinded treatment for a variable duration beyond 52 weeks.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment sequence if any of the entry criteria were violated.
Groups:
- Placebo: Participants received placebo matching 9 mg or 18 mg nerandomilast film coated tablet orally twice daily, with doses given at least 12 hours apart and each taken with 250 mL of water.
Period: Overall Study
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Started (Started Trial Medication) | 393 | 392 | 392
Completed Treatment Period A (52 Weeks) | 320 | 324 | 318
Completed (Completed planned trial treatment period over the whole trial) | 292 | 298 | 299
Not Completed | 101 | 94 | 93
Not completed — Adverse Event | 52 | 52 | 64
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 23 | 18 | 12
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — No reason stated by the participants | 23 | 22 | 16
Not completed — Lack of Efficacy | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo matching 9 mg or 18 mg nerandomilast orally twice daily, with doses given at least 12 hours apart and each taken with 250 mL of water.
- Total: Total of all reporting groups
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID | Total
Number analyzed (Participants) | 393 | 392 | 392 | 1177
Age, Continuous [Mean (Standard Deviation); unit: Years] — Full Analysis Set (FAS):
  This patient set includes all randomized patients who received at least one dose of study drug.
  Years | 69.9 (7.5) | 70.5 (7.8) | 70.3 (7.8) | 70.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
  Participants
    Female | 56 | 75 | 69 | 200
    Male | 337 | 317 | 323 | 977
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
  Participants
    Hispanic or Latino | 28 | 23 | 44 | 95
    Not Hispanic or Latino | 365 | 369 | 348 | 1082
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
  Participants
    American Indian or Alaska Native | 1 | 2 | 2 | 5
    Asian | 116 | 121 | 130 | 367
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 2 | 3 | 1 | 6
    White | 273 | 266 | 258 | 797
    More than one race | 1 | 0 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0
Forced Vital Capacity (FVC) at baseline [Mean (Standard Deviation); unit: Milliliters (mL)] — Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
  Milliliters (mL) | 2863.9 (804.6) | 2837.2 (781.4) | 2827.3 (758.0) | 2842.8 (781.1)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC) [mL] at Week 52
Description: The absolute change from baseline in Forced Vital Capacity (FVC) [mL] at Week 52 is reported.
  The absolute change from baseline in forced vital capacity (FVC) at Week 52 was analyzed using a restricted maximum likelihood (REML)-based mixed model with repeated measures (MMRM). The model included fixed categorical effects of treatment and baseline antifibrotic use at each visit, as well as the continuous effect of baseline FVC. Visit was treated as a repeated measure, with an unstructured covariance structure for within-patient variability.
Time Frame: The MMRM model is a longitudinal analysis, and it incorporated FVC measurements from baseline (Week -8 to Week -1) and Week 2, Week 6, Week 12, Week 18, Week 26, Week 36, Week 44 and Week 52. The data represent the Least Squares Mean at Week 52
Population: Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug. only patients with baseline measurement and at least one post-baseline measurement are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliliters (mL)
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 391 | 390 | 392
Milliliters (mL) | -183.48 [-210.86 to -156.10] | -138.60 [-165.59 to -111.61] | -114.65 [-141.81 to -87.50]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; Based on a Mixed Model for Repeated Measures (MMRM), which included fixed, categorical effects of treatment at each visit, baseline use of antifibrotic therapy at each visit, and fixed continuous effects of baseline forced vital capacity (FVC) in milliliters at each visit. Patients were treated as a random effect. Visit was treated as the repeated measure, and an unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p = 0.0222, Mixed Models Analysis; The Kenward-Roger method estimated denominator degrees of freedom and adjusted standard errors; tests used two-sided α per multiple testing strategy; Mean Difference (Net) = 44.89, 95% CI 2-sided [6.44 to 83.33] — Adjusted mean difference in FVC change from baseline at Week 52 between the Nera 9 mg bid group and the Placebo group
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 68.83, 95% CI 2-sided [30.26 to 107.39] — Adjusted mean difference in FVC change from baseline at Week 52 between the Nera 18 mg bid group and the Placebo group

2. Secondary Outcome: Key Secondary Endpoint: Time to the First Occurrence of Any of the Components of the Composite Endpoint: Time to First Acute IPF Exacerbation, First Hospitalization for Respiratory Cause, or Death (Whichever Occurs First) Over the Duration of the Trial
Description: Time to the first occurrence of any component of the composite endpoint-acute IPF exacerbation, hospitalization for a respiratory cause, or death (whichever occurred first)-is reported as the number of participants who experienced one or more of these events during the trial.
  Acute IPF is defined as an acute, clinically significant respiratory deterioration characterized by evidence of new, widespread alveolar abnormality, with all of the following:
  Acute worsening or development of dyspnea, typically of less than 1 month's duration.
  Computed tomography showing new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with IPF.
  Deterioration not fully explained by cardiac failure or fluid overload.
  If more than one component occurred on the same day, the patient was counted under the first event according to the following hierarchy: acute IPF exacerbation, hospitalization, death.
Time Frame: From first administration of any trial drug (Nerandomilast or Placebo) up to 22.9 months.
Population: Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 393 | 392 | 392
Participants
  Acute IPF exacerbation as the first event | 38 | 32 | 38
  Hospitalisation for respiratory cause as the first event | 49 | 45 | 47
  Death as the first event | 16 | 13 | 8
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; The hazard ratio (HR) was estimated using a Cox proportional hazards model with treatment group, baseline antifibrotic therapy use, age (continuous), baseline FVC % predicted, and baseline DLCO % predicted (hemoglobin-corrected) as covariates. Breslow's method was applied for tied event times. A two-sided p-value from the Wald test assessed the treatment effect. P-values were not adjusted for multiplicity; Test type: Superiority; p = 0.5443, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.69 to 1.22]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; Based on Cox proportional hazards model including treatment, baseline antifibrotic therapy, age, baseline Forced Vital Capacity (FVC) percent predicted, and baseline Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) percent predicted (corrected for haemoglobin) as covariates. p-values not adjusted for multiplicity; Test type: Superiority; p = 0.9512, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.75 to 1.31]

3. Secondary Outcome: Time to First Acute IPF Exacerbation or Death Over the Duration of the Trial
Description: The time to first acute IPF exacerbation or death during the trial is reported as the number of participants who experienced either event.
  Acute IPF is defined as an acute, clinically significant respiratory deterioration characterized by evidence of new, widespread alveolar abnormality, with all of the following:
  Acute worsening or development of dyspnea, typically of less than 1 month's duration.
  Computed tomography showing new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with IPF.
  Deterioration not fully explained by cardiac failure or fluid overload.
  If more than one component occurred on the same day, the patient was counted under the first event according to the following hierarchy: acute IPF exacerbation followed by death.
Time Frame: From first administration of any trial drug (Nerandomilast or Placebo) up to 22.9 months.
Population: Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 393 | 392 | 392
Participants
  Acute IPF exacerbation | 30 | 31 | 38
  Death | 19 | 20 | 12
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; Analysis was performed using a Cox proportional hazards regression model that included baseline use of antifibrotic therapy (antifibrotic group vs non-antifibrotic group), age, baseline forced vital capacity (FVC) percentage predicted, baseline diffusing capacity of the lungs for carbon monoxide (DLCO) percentage predicted (corrected for hemoglobin levels), and treatment group as covariates; Test type: Superiority; p = 0.5583, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.76 to 1.67]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5896, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.75 to 1.65]

4. Secondary Outcome: Time to Hospitalization for Respiratory Cause or Death Over the Duration of the Trial
Description: Time to hospitalization for respiratory cause or death over the duration of the trial is reported as the number of participants who experienced either event.
  Hospitalizations due to respiratory causes were recorded on a specific non-elective hospitalization CRF page. This page captured the hospitalization date, confirmation of a respiratory cause, and the primary admission diagnosis.
  If more than one component occurred on the same day, the patient was counted under the first event according to the hierarchy: hospitalization for respiratory cause, followed by death.
Time Frame: From first administration of any trial drug (Nerandomilast or Placebo) up to 22.9 months.
Population: Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 393 | 392 | 392
Participants
  Hospitalization for respiratory cause | 59 | 57 | 68
  Death | 14 | 11 | 7
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9038, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.70 to 1.36]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4687, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.82 to 1.56]

5. Secondary Outcome: Time to Absolute Decline in Forced Vital Capacity (FVC) % Predicted of >10% From Baseline or Death Over the Duration of the Trial
Description: The time to absolute decline of more than 10% from baseline in forced vital capacity (FVC) percent predicted, or death, over the duration of the trial is reported as the number of participants who experienced either event.
  If more than one component occurred on the same day, the patient was counted under the first event according to the hierarchy; Absolute decline in FVC % predicted of > 10% followed by death.
Time Frame: From first administration of any trial drug (Nerandomilast or Placebo) up to 22.9 months.
Population: Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 393 | 392 | 392
Participants
  Absolute decline in FVC % predicted of > 10% | 91 | 89 | 80
  Death | 20 | 18 | 14
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.7695, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.74 to 1.25]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2068, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.64 to 1.10]

6. Secondary Outcome: Time to Absolute Decline in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) Percentage Predicted by More Than 15% From Baseline or Death, Measured Over the Duration of the Trial
Description: The time to absolute decline of more than 15% from baseline in diffusing capacity of the lungs for carbon monoxide (DLCO) percent predicted, or death, over the duration of the trial is reported as the number of participants who experienced either event.
  Predicted DLCO value was corrected for hemoglobin (Hb).
  If more than one component occurred on the same day, the patient was counted under the first event according to the hierarchy: Absolute decline in DLCO % predicted of > 15%, followed by Death.
Time Frame: From first administration of any trial drug (Nerandomilast or Placebo) up to 22.9 months.
Population: Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 393 | 392 | 392
Participants
  Absolute decline in DLCO % predicted of > 15% | 38 | 35 | 43
  Death | 28 | 24 | 16
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9251, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.69 to 1.41]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4988, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.62 to 1.26]

7. Secondary Outcome: Time to Death Over the Duration of the Trial
Description: Time to death over the duration of the trial is reported as the number of participants who died.
  Time to death will be based either on the date of death on the AE report for patients with AEs leading to death or will be based on the information from the vital status assessment.
Time Frame: From first administration of any trial drug (Nerandomilast or Placebo) up to 22.9 months.
Population: Full Analysis Set (FAS): This patient set includes all randomized patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 393 | 392 | 392
Participants | 28 | 26 | 21
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9084, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.60 to 1.76]
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4682, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.46 to 1.43]

8. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Symptoms Dyspnea Domain Score at Week 52
Description: The absolute change from baseline in the Living with Pulmonary Fibrosis (L-PF) Symptoms Dyspnea domain score at Week 52 is reported. This endpoint was analyzed using a Mixed Model for Repeated Measures (MMRM). The model included fixed effects for treatment, baseline use of antifibrotic therapy, and baseline dyspnea score at each visit, with an unstructured covariance structure to model repeated measures.
  The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44-item tool consisting of two modules:
  Symptoms (23 items) and
  Impacts (21 items).
  The Symptoms module yields three domain scores:
  Dyspnea,
  Cough, and
  Fatigue,
  as well as a Total Symptoms score.
  Scoring is based on the mean of item ratings within each domain, multiplied by 100.
  Scores range from 0 to 100, with higher scores indicating greater impairment.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated L-PF measurements from baseline (Week -8 to Week -1) and Week 12, Week 26, Week 36, Week 44 and Week 52. The data represent the Least Squares Mean at Week 52.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 380 | 375 | 385
Score on a scale | 7.26 [5.70 to 8.82] | 6.26 [4.71 to 7.80] | 6.63 [5.09 to 8.17]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; The analysis used a Mixed Model for Repeated Measures (MMRM) with fixed categorical effects for treatment group and baseline antifibrotic therapy at each visit, and fixed continuous effects of baseline Living with Pulmonary Fibrosis (L-PF) Dyspnea domain score. An unstructured covariance structure accounted for within-patient correlations. Baseline antifibrotic use, as recorded in the concomitant medication case report form (CRF), was included as a covariate; Test type: Superiority; p = 0.3697, Mixed Models Analysis; Mean Difference (Net) = -1.00, 95% CI 2-sided [-3.20 to 1.19] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Dyspnea score) between the Nera 9mg BID group and the Placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.5734, Mixed Models Analysis; Mean Difference (Net) = -0.63, 95% CI 2-sided [-2.83 to 1.57] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Dyspnea score) between the Nera 18mg BID group and the Placebo group at Week 52

9. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Symptoms Cough Domain Score at Week 52
Description: The absolute change from baseline in the L-PF Cough domain score at Week 52 is reported. This endpoint was analyzed using a Mixed Model for Repeated Measures (MMRM). The model included fixed effects for treatment, baseline antifibrotic therapy, and baseline L-PF Cough score at each visit, with an unstructured covariance matrix for repeated measures.
  The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44-item tool consisting of two modules:
  Symptoms (23 items) and
  Impacts (21 items).
  The Symptoms module yields three domain scores:
  Dyspnea,
  Cough, and
  Fatigue,
  as well as a Total Symptoms score.
  Scoring is based on the mean of item ratings within each domain, multiplied by 100.
  Scores range from 0 to 100, with higher scores indicating greater impairment.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 379 | 373 | 385
Score on a scale | 4.54 [2.49 to 6.59] | 4.44 [2.42 to 6.46] | 3.95 [1.93 to 5.97]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; The analysis was based on a Mixed Model for Repeated Measures (MMRM), which included fixed categorical effects for treatment group at each visit, baseline use of antifibrotic therapy at each visit, and fixed continuous effects of the baseline Living with Pulmonary Fibrosis (L-PF) Cough domain score at each visit. An unstructured covariance structure modeled repeated measures. Baseline antifibrotic use, recorded in the concomitant medication case report form (CRF), was included as a covariate; Test type: Superiority; p = 0.9442, Mixed Models Analysis; Mean Difference (Net) = -0.10, 95% CI 2-sided [-2.98 to 2.77] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Cough score) between the Nera 9 mg BID group and the Placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.6862, Mixed Models Analysis; Mean Difference (Net) = -0.59, 95% CI 2-sided [-3.47 to 2.28] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Cough score) between the Nera 18 mg BID group and the Placebo group at Week 52

10. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Symptoms Fatigue Domain Score at Week 52
Description: The absolute change from baseline in the Living with Pulmonary Fibrosis (L-PF) Fatigue domain score at Week 52 is reported.
  The analysis used a mixed model for repeated measures (MMRM) with fixed categorical effects for treatment, baseline antifibrotic (AF) therapy, and the fixed continuous effect of baseline L-PF score. Covariance was unstructured. Baseline AF therapy was a covariate.
  The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44-item tool consisting of two modules:
  Symptoms (23 items) and
  Impacts (21 items).
  The Symptoms module yields three domain scores:
  Dyspnea,
  Cough, and
  Fatigue,
  as well as a Total Symptoms score.
  Scoring is based on the mean of item ratings within each domain, multiplied by 100.
  Scores range from 0 to 100, with higher scores indicating greater impairment.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 380 | 375 | 386
Score on a scale | 5.40 [3.66 to 7.14] | 5.59 [3.88 to 7.30] | 5.82 [4.11 to 7.54]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; The analysis was based on a Mixed Model for Repeated Measures (MMRM), which included fixed categorical effects for treatment group at each visit, baseline use of antifibrotic therapy at each visit, and fixed continuous effects of the baseline Living with Pulmonary Fibrosis (L-PF) Fatigue domain score at each visit. An unstructured covariance structure modeled repeated measures. Baseline antifibrotic use, recorded in the concomitant medication case report form (CRF), was included as a covariate; Test type: Superiority; p = 0.8759, Mixed Models Analysis; Mean Difference (Net) = 0.19, 95% CI 2-sided [-2.25 to 2.63] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Fatigue score) between the Nera 9 mg BID group and the Placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.7320, Mixed Models Analysis; Mean Difference (Net) = 0.43, 95% CI 2-sided [-2.02 to 2.87] — The adjusted mean difference represents the model-estimated difference in symptom change (L-PF Fatigue score) between the Nera 18 mg BID group and the Placebo group at Week 52

11. Secondary Outcome: Absolute Change From Baseline in Forced Vital Capacity Percent Predicted at Week 52
Description: The absolute change from baseline in Forced Vital Capacity percent predicted at Week 52 is reported.
  Analysis was based on a Mixed Model for Repeated Measures (MMRM), which included fixed, categorical effects of treatment at each visit, baseline use of antifibrotic therapy at each visit, and the fixed continuous effects of baseline forced vital capacity (FVC) percentage predicted at each visit. An unstructured covariance structure was used to model repeated measures within patients.
  Baseline use of antifibrotic therapy, as recorded in the concomitant medication case report form (CRF) page, was included as a covariate.
Time Frame: The MMRM model is a longitudinal analysis, and it incorporated FVC measurements from baseline (Week -8 to Week -1) and Week 1, Week 2, Week 6, Week 12, Week 18, Week 26, Week 36, Week 44 and Week 52. The data represent the Least Squares Mean at Week 52.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: FVC percent predicted
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 391 | 390 | 392
FVC percent predicted | -4.92 [-5.67 to -4.18] | -3.75 [-4.48 to -3.01] | -3.19 [-3.93 to -2.45]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; Analysis was based on a Mixed Model for Repeated Measures (MMRM), which included fixed, categorical effects of treatment, baseline use of antifibrotic therapy, and the fixed continuous effects of baseline forced vital capacity (FVC) percentage predicted at each visit. An unstructured covariance structure was used to model repeated measures within patients. Baseline use of antifibrotic therapy, as recorded in the concomitant medication case report form (CRF) page, was included as a covariate; Test type: Superiority; p = 0.0280, Mixed Models Analysis; Mean Difference (Net) = 1.17, 95% CI 2-sided [0.13 to 2.22] — The adjusted mean difference represents the model-estimated difference in percent predicted Forced Vital Capacity between the Nera 9 mg BID group and the placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0013, Mixed Models Analysis; Mean Difference (Net) = 1.73, 95% CI 2-sided [0.68 to 2.78] — The adjusted mean difference represents the model-estimated difference in percent predicted Forced Vital Capacity between the Nera 18 mg BID group and the placebo group at Week 52

12. Secondary Outcome: Absolute Change From Baseline in Diffusing Capacity of the Lungs for Carbon Monoxide Percent Predicted at Week 52
Description: The absolute change from baseline in Diffusing Capacity of the Lungs for Carbon Monoxide percent predicted at Week 52 is reported.
  The analysis was based on a Mixed Model for Repeated Measures (MMRM), which included fixed, categorical effects of treatment at each visit, baseline use of antifibrotic therapy at each visit, and the fixed continuous effects of baseline diffusing capacity of the lungs for carbon monoxide (DLCO) percentage predicted at each visit. An unstructured covariance structure was used to model repeated measures within patients.
  Baseline use of antifibrotic therapy, as recorded in the concomitant medication case report form (CRF) page, was included as a covariate.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated DLCO measurements from baseline (Week -8 to Week -1) and Week 12, Week 26, and Week 52. The data represent the Least Squares Mean at Week 52.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: DLCO percent predicted
Arm/Group | Placebo | Nerandomilast 9 mg BID | Nerandomilast 18 mg BID
Number analyzed (Participants) | 380 | 378 | 384
DLCO percent predicted | -6.14 [-7.35 to -4.94] | -3.66 [-4.85 to -2.46] | -4.47 [-5.66 to -3.27]
Statistical Analysis 1: Comparison: Placebo vs Nerandomilast 9 mg BID; Based on a Mixed Model for Repeated Measures (MMRM), which included fixed, categorical effects of treatment, baseline use of antifibrotic therapy, and the fixed continuous effects of baseline diffusing capacity of the lungs for carbon monoxide (DLCO) percentage predicted at each visit. An unstructured covariance structure was used to model repeated measures within patients. Baseline use of antifibrotic therapy, as recorded in the concomitant medication CRF page, was included as a covariate; Test type: Superiority; p = 0.0042, Mixed Models Analysis; Mean Difference (Net) = 2.49, 95% CI 2-sided [0.79 to 4.19] — The adjusted mean difference represents the model-estimated difference in percent predicted DLCO between the Nera 9 mg BID group and the placebo group at Week 52
Statistical Analysis 2: Comparison: Placebo vs Nerandomilast 18 mg BID; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0530, Mixed Models Analysis; Mean Difference (Net) = 1.67, 95% CI 2-sided [-0.02 to 3.37] — The adjusted mean difference represents the model-estimated difference in percent predicted DLCO between the Nera 18 mg BID group and the placebo group at Week 52

ADVERSE EVENTS:
Time Frame: AE collection and All-cause mortality From first trial drug administration (Placebo or Nerandomilast) up to 22.9 months.
Description: Treated Set (TS): This patient set includes all randomized patients who received at least one dose of study drug.
Groups:
- Nera 9 mg BID: Participants received 9 mg film-coated nerandomilast tablets orally twice daily, with doses administered at least 12 hours apart, each taken with 250 mL of water.
- Nera 18 mg BID: Participants received 18 mg film-coated nerandomilast tablets orally twice daily, with doses administered at least 12 hours apart, each taken with 250 mL of water.
Arm/Group | Placebo | Nera 9 mg BID | Nera 18 mg BID
All-Cause Mortality (participants affected / at risk) | 42/393 | 36/392 | 26/392
Serious Adverse Events (participants affected / at risk) | 181/393 | 159/392 | 165/392
Other Adverse Events (participants affected / at risk) | 316/393 | 319/392 | 337/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=393) | Nera 9 mg BID (N=392) | Nera 18 mg BID (N=392)
Acquired factor VIII deficiency (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 3 | 2
Acute right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 2 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3
Atrial flutter (Cardiac disorders) | 2 | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 3 | 1
Cardiac failure (Cardiac disorders) | 3 | 1 | 5
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0
Cor pulmonale chronic (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 2
Coronary artery dissection (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1
Heart failure with preserved ejection fraction (Cardiac disorders) | 1 | 1 | 0
Heart failure with reduced ejection fraction (Cardiac disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 2 | 0
Left ventricular failure (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 3 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1
Retinopathy congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1
Presbyacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 1
Amaurosis (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 2 | 0 | 2
Dry age-related macular degeneration (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Hypotony of eye (Eye disorders) | 1 | 0 | 0
Retinal infarction (Eye disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 1 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 3
Intestinal mass (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Oronasal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 1 | 1 | 3
Chest pain (General disorders) | 2 | 3 | 0
Condition aggravated (General disorders) | 34 | 28 | 32
Death (General disorders) | 5 | 4 | 2
Disease progression (General disorders) | 2 | 0 | 3
Gait disturbance (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 1
Illness (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 2
Sudden death (General disorders) | 1 | 0 | 0
Vascular stent stenosis (General disorders) | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Suspected drug-induced liver injury (Hepatobiliary disorders) | 2 | 1 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Appendiceal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1
Aspergillus infection (Infections and infestations) | 0 | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 2
Biliary tract infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 2
COVID-19 (Infections and infestations) | 2 | 4 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 1 | 0 | 0
HCoV-OC43 infection (Infections and infestations) | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 3 | 3 | 2
Laryngitis (Infections and infestations) | 2 | 0 | 0
Latent tuberculosis (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 1
Pleurisy bacterial (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 22 | 18 | 17
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 6 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1 | 4
Salmonellosis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3
Urinary tract infection (Infections and infestations) | 3 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Venomous bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 2
Clostridium test positive (Investigations) | 0 | 0 | 1
False positive investigation result (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1
Influenza A virus test positive (Investigations) | 1 | 0 | 0
Interferon gamma release assay positive (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 1
Queyrat erythroplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sarcomatoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 1
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Carotid artery dissection (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 2
Dementia (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 1
Focal dyscognitive seizures (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Middle cerebral artery stroke (Nervous system disorders) | 0 | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 1 | 0 | 0
Subdural hygroma (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 3 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0
Hallucinations, mixed (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 3 | 3
Tobacco abuse (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 5 | 3
Nephritis (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 12 | 13 | 11
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 8
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 12
Pulmonary venous hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 4
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Assisted suicide (Surgical and medical procedures) | 0 | 1 | 0
Aneurysm (Vascular disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 1 | 0
Aortic dilatation (Vascular disorders) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 1
Granulomatosis with polyangiitis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 0
Microscopic polyangiitis (Vascular disorders) | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1 | 3
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=393) | Nera 9 mg BID (N=392) | Nera 18 mg BID (N=392)
Diarrhoea (Gastrointestinal disorders) | 75 | 130 | 166
Nausea (Gastrointestinal disorders) | 28 | 39 | 33
Vomiting (Gastrointestinal disorders) | 19 | 19 | 21
Condition aggravated (General disorders) | 27 | 19 | 27
Fatigue (General disorders) | 23 | 35 | 30
Bronchitis (Infections and infestations) | 37 | 35 | 37
COVID-19 (Infections and infestations) | 61 | 74 | 59
Nasopharyngitis (Infections and infestations) | 53 | 46 | 49
Pneumonia (Infections and infestations) | 17 | 21 | 18
Respiratory tract infection (Infections and infestations) | 12 | 15 | 23
Upper respiratory tract infection (Infections and infestations) | 47 | 49 | 56
Weight decreased (Investigations) | 39 | 45 | 54
Decreased appetite (Metabolism and nutrition disorders) | 28 | 39 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 23 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 25 | 31
Dizziness (Nervous system disorders) | 21 | 28 | 19
Headache (Nervous system disorders) | 23 | 27 | 28
Anxiety (Psychiatric disorders) | 40 | 35 | 44
Depression (Psychiatric disorders) | 38 | 42 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 79 | 74 | 73
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 58 | 50 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT05321069/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT05321069/SAP_001.pdf